CLINICAL TRIAL: NCT03335644
Title: The NutriNet-Santé Study. A Web-based Prospective Cohort Study of the Relationship Between Nutrition and Health and of Dietary Patterns and Nutritional Status Predictors
Brief Title: The NutriNet-Santé Study
Status: Recruiting | Type: Observational
Sponsor: University of Paris 13 (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Conservatoire national des Arts et Métiers (Other)
Responsible Party: Principal Investigator, Mathilde Touvier, Dr, University of Paris 13
Other Study IDs: NutriNet-Santé
Record Dates: First submitted 2017-10-11; First posted 2017-11-08 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Diet, Food, and Nutrition; Exercise; Diseases Category; Cohort Studies; Adult; Anthropometry; Humans; Internet; Surveys and Questionnaires; Mortality
Keywords: determinants of dietary patterns and nutritional status; Food additives, Food processing; Exclusion diets, vegetarian diet, vegan diet; Organic food, pesticide exposure, sustainability; Gut microbiota; Food labeling; Dietary supplements; Food based dietary guidelines; Psychological determinants of food behavior; Geographical determinants of food behavior; Breastfeeding; Mental health; Cancer; Cardiovascular and cardiometabolic health; Multimorbidity
MeSH Terms: conditions — Motor Activity; Breast Feeding; Psychological Well-Being; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of serum, plasma, and buffy-coats (for genetic analyses), as well as urine samples was set up for 19 600 subjects of the cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NutriNet-Santé study was set up to investigate nutrition and health relationships. Specifically, it was the first web-based cohort worldwide on such a large scale (n=171 000 as of 2021) focused on the complex link between nutrition and health status. It is characterized by a very detailed assessment of nutritional exposure and dietary behavior.

https://etude-nutrinet-sante.fr/ https://info.etude-nutrinet-sante.fr/en

DETAILED DESCRIPTION:
NutriNet-Santé is a large-scale (n=171,000) web-based cohort coordinated by EREN, launched in France in 2009 to investigate nutrition and health relationships. All required ethics authorisations have been obtained (listed here). NutriNet-Santé participants regularly fill questionnaires through a dedicated and secure website, providing extensive, high-quality nutritional and non-nutritional data, including repeated data on socio-demographics and lifestyle (yearly), anthropometrics (every 6 months), dietary intake (every 6 months), physical activity (IPAQ questionnaire, yearly)5 and health status (every 6 months). NutriNet-Santé is characterised by a very detailed and up-to-date assessment of nutritional exposure and dietary behaviours. Usual dietary intakes are assessed at baseline and every 6 months thereafter through a series of 3 non-consecutive randomly assigned 24h dietary records. Daily energy, alcohol, micro- and macronutrient intakes are calculated using the published NutriNet-Santé food composition database (>3,500 generic items). All major health events (e.g., cancers, cardio- and cerebrovascular diseases) are reported by the participants and validated by an expert committee of physicians based on medical records, and/or retrieved from the French National Health Insurance medico-administrative databases to limit potential reporting bias. In turn, mortality data are obtained from the exhaustive French National Mortality Registry (CépiDC). The number of incident events already registered is as follows: 4,200 cancers and 1,240 deaths. A sub-sample of the cohort (n=20,000) provided blood and urine samples, currently stored at -80°C in EREN's biobank.

ELIGIBILITY:
Inclusion Criteria:

* aged over 15 years
* access to internet

Exclusion Criteria:

* aged under 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The NutriNet-Santé study is a French ongoing web-based cohort launched in 2009 with the objective to study the associations between nutrition and health as well as the determinants of dietary behaviors and nutritional status. This cohort has been previously described in details (citations). Participants aged over 15 years with access to the Internet are recruited by vast multimedia campaigns. All questionnaires are completed online using a dedicated website (www.etude-nutrinet-sante.fr).
Sampling Method: Non-Probability Sample
Enrollment: 170000 (Estimated)
Dates: Start 2009-05-11 (Actual); Primary Completion 2029-05-11 (Estimated); Study Completion 2029-05-11 (Estimated)

PRIMARY OUTCOMES:
cancers using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
CVD using health questionnaire and/or the dedicated website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
type 2 diabetes using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
hypertension using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
metabolic syndrome using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
depression using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
migraine using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
rheumatoid arthritis using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
cognitive decline using health questionnaire and/or the website for declaration of major health events | every 6 months after registration, up to 10 years of follow-up
  self reported
quality of life using the SF-36 questionnaire | every 6 months after registration, up to 10 years of follow-up
  self reported
Weight using anthropometric questionnaire | every year after registration, up to 10 years of follow-up
  self reported
Height using anthropometric questionnaire | every year after registration, up to 10 years of follow-up
  self reported
Mortality | continuously updated
  CepiDC exhaustive national registry
Mental health (incl. anxious disorders, sleep disorders, addictive behaviors, eating disorders) | repeatedly during followup
  self reported though validated scales and/or questionnaires
SARSCOV-2 (Covid 19) infection | regular update for a subsampe of the cohort from 2020
  serology + questionnaires on symptoms
multi-morbidity (mental and physical health) | continuous update
  combination of previsously listed mental and physical health outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- EREN, Bobigny, Seine Saint Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hercberg S, Castetbon K, Czernichow S, Malon A, Mejean C, Kesse E, Touvier M, Galan P. The Nutrinet-Sante Study: a web-based prospective study on the relationship between nutrition and health and determinants of dietary patterns and nutritional status. BMC Public Health. 2010 May 11;10:242. doi: 10.1186/1471-2458-10-242. PMID 20459807
- [Derived] Hasenbohler A, Javaux G, Payen de la Garanderie M, Szabo de Edelenyi F, Bourhis L, Agaesse C, De Sa A, Huybrechts I, Pierre F, Coumoul X, Julia C, Kesse-Guyot E, Alles B, Fezeu LK, Hercberg S, Deschasaux-Tanguy M, Cosson E, Tatulashvili S, Chassaing B, Srour B, Touvier M. Associations between preservative food additives and type 2 diabetes incidence in the NutriNet-Sante prospective cohort. Nat Commun. 2026 Jan 7;16(1):11199. doi: 10.1038/s41467-025-67360-w. PMID 41501013
- [Derived] Hasenbohler A, Javaux G, Payen de la Garanderie M, de Edelenyi FS, Yvroud-Hoyos P, Agaesse C, De Sa A, Huybrechts I, Pierre F, Audebert M, Coumoul X, Julia C, Kesse-Guyot E, Alles B, Deschamps V, Hercberg S, Chassaing B, Srour B, Deschasaux-Tanguy M, Touvier M. Intake of food additive preservatives and incidence of cancer: results from the NutriNet-Sante prospective cohort. BMJ. 2026 Jan 7;392:e084917. doi: 10.1136/bmj-2025-084917. PMID 41500678
- [Derived] Cote M, Hutchinson JM, Touvier M, Srour B, Bourhis L, Lamarche B, Fezeu LK. Associations between Dietary Pattern Networks Derived from Machine Learning Algorithms and Cardiovascular Disease Risk in the NutriNet-Sante Cohort. J Nutr. 2025 Nov;155(11):4033-4042. doi: 10.1016/j.tjnut.2025.09.014. Epub 2025 Sep 22. PMID 40992665
- [Derived] Paz-Graniel I, Kose J, Duquenne P, Babio N, Salas-Salvado J, Hercberg S, Galan P, Touvier M, Fezeu LK, Andreeva VA. Alcohol, Smoking, and Their Synergy as Risk Factors for Incident Type 2 Diabetes. Am J Prev Med. 2025 Nov;69(5):108011. doi: 10.1016/j.amepre.2025.108011. Epub 2025 Jul 31. PMID 40752888
- [Derived] Berthy F, Toujgani H, Duquenne P, Fezeu LK, Lairon D, Pointereau P, Touvier M, Hercberg S, Galan P, Alles B, Baudry J, Kesse-Guyot E. Prospective association of the EAT-Lancet reference diet with body weight changes and incidence of overweight and obesity in a French cohort. Am J Clin Nutr. 2025 Aug;122(2):450-459. doi: 10.1016/j.ajcnut.2025.06.013. Epub 2025 Jun 17. PMID 40553762
- [Derived] Toujgani H, Wang J, Perraud E, Baudry J, Berlivet J, Alles B, Fouillet H, Hercberg S, Touvier M, Lairon D, Pointereau P, Couturier C, Mariotti F, Kesse-Guyot E; TRANSFood Consortium. Dietary consumption trajectory profiles over time of French adults from the NutriNet-Sante cohort (2014-2022): multicriteria analysis of sustainability. Int J Behav Nutr Phys Act. 2025 Jun 13;22(1):76. doi: 10.1186/s12966-025-01777-w. PMID 40514663
- [Derived] Paolassini-Guesnier P, Van Beekum M, Kesse-Guyot E, Baudry J, Shankland R, Rodhain A, Bellicha A, Leys C, Hercberg S, Touvier M, Alles B, Peneau S. Mindful eating is associated with a healthier plant-based diet in the NutriNet-Sante study. Sci Rep. 2025 Jun 6;15(1):19928. doi: 10.1038/s41598-025-02195-5. PMID 40481021
- [Derived] Meyer E, Alles B, Berlivet J, Peneau S, Bellicha A, Touvier M, Langevin B, Pointereau P, Lairon D, Hercberg S, Kesse-Guyot E, Baudry J. Typology of out-of-home eaters: a description of sociodemographic, lifestyle, nutritional and environmental characteristics in the NutriNet-Sante cohort. Int J Behav Nutr Phys Act. 2025 May 26;22(1):61. doi: 10.1186/s12966-025-01752-5. PMID 40420193
- [Derived] Payen de la Garanderie M, Hasenbohler A, Dechamp N, Javaux G, Szabo de Edelenyi F, Agaesse C, De Sa A, Bourhis L, Porcher R, Pierre F, Coumoul X, Kesse-Guyot E, Alles B, Fezeu LK, Cosson E, Tatulashvili S, Huybrechts I, Hercberg S, Deschasaux-Tanguy M, Chassaing B, Rytter H, Srour B, Touvier M. Food additive mixtures and type 2 diabetes incidence: Results from the NutriNet-Sante prospective cohort. PLoS Med. 2025 Apr 8;22(4):e1004570. doi: 10.1371/journal.pmed.1004570. eCollection 2025 Apr. PMID 40198579
- [Derived] Gomez-Martinez C, Paolassini-Guesnier P, Fezeu L, Srour B, Hercberg S, Touvier M, Babio N, Salas-Salvado J, Peneau S. Trait impulsivity is associated with an increased risk of type 2 diabetes incidence in adults over 8 years of follow-up: results from the NutriNet-Sante cohort. BMC Med. 2024 Aug 15;22(1):332. doi: 10.1186/s12916-024-03540-7. PMID 39148083
- [Derived] Salame C, Javaux G, Sellem L, Viennois E, de Edelenyi FS, Agaesse C, De Sa A, Huybrechts I, Pierre F, Coumoul X, Julia C, Kesse-Guyot E, Alles B, Fezeu LK, Hercberg S, Deschasaux-Tanguy M, Cosson E, Tatulashvili S, Chassaing B, Srour B, Touvier M. Food additive emulsifiers and the risk of type 2 diabetes: analysis of data from the NutriNet-Sante prospective cohort study. Lancet Diabetes Endocrinol. 2024 May;12(5):339-349. doi: 10.1016/S2213-8587(24)00086-X. PMID 38663950
- [Derived] Duquenne P, Capperella J, Fezeu LK, Srour B, Benasi G, Hercberg S, Touvier M, Andreeva VA, St-Onge MP. The Association Between Ultra-Processed Food Consumption and Chronic Insomnia in the NutriNet-Sante Study. J Acad Nutr Diet. 2024 Sep;124(9):1109-1117.e2. doi: 10.1016/j.jand.2024.02.015. Epub 2024 Feb 28. PMID 38423510
- [Derived] Sellem L, Srour B, Javaux G, Chazelas E, Chassaing B, Viennois E, Debras C, Druesne-Pecollo N, Esseddik Y, Szabo de Edelenyi F, Arnault N, Agaesse C, De Sa A, Lutchia R, Huybrechts I, Scalbert A, Pierre F, Coumoul X, Julia C, Kesse-Guyot E, Alles B, Galan P, Hercberg S, Deschasaux-Tanguy M, Touvier M. Food additive emulsifiers and cancer risk: Results from the French prospective NutriNet-Sante cohort. PLoS Med. 2024 Feb 13;21(2):e1004338. doi: 10.1371/journal.pmed.1004338. eCollection 2024 Feb. PMID 38349899
- [Derived] Reuze A, Mejean C, Sirieix L, Baudry J, Kesse-Guyot E, Druesne-Pecollo N, Brunin J, Hercberg S, Touvier M, Peneau S, Alles B. Stages of Change toward Meat Reduction: Associations with Motives and Longitudinal Dietary Data on Animal-Based and Plant-Based Food Intakes in French Adults. J Nutr. 2023 Nov;153(11):3295-3307. doi: 10.1016/j.tjnut.2023.09.017. Epub 2023 Sep 28. PMID 37774842
- [Derived] Sellem L, Srour B, Javaux G, Chazelas E, Chassaing B, Viennois E, Debras C, Salame C, Druesne-Pecollo N, Esseddik Y, de Edelenyi FS, Agaesse C, De Sa A, Lutchia R, Louveau E, Huybrechts I, Pierre F, Coumoul X, Fezeu LK, Julia C, Kesse-Guyot E, Alles B, Galan P, Hercberg S, Deschasaux-Tanguy M, Touvier M. Food additive emulsifiers and risk of cardiovascular disease in the NutriNet-Sante cohort: prospective cohort study. BMJ. 2023 Sep 6;382:e076058. doi: 10.1136/bmj-2023-076058. PMID 37673430
- [Derived] Berthy F, Brunin J, Alles B, Reuze A, Touvier M, Hercberg S, Lairon D, Pointereau P, Mariotti F, Baudry J, Kesse-Guyot E. Higher adherence to the EAT-Lancet reference diet is associated with higher nutrient adequacy in the NutriNet-Sante cohort: a cross-sectional study. Am J Clin Nutr. 2023 Jun;117(6):1174-1185. doi: 10.1016/j.ajcnut.2023.03.029. Epub 2023 Apr 3. PMID 37019361
- [Derived] Srour B, Chazelas E, Druesne-Pecollo N, Esseddik Y, de Edelenyi FS, Agaesse C, De Sa A, Lutchia R, Debras C, Sellem L, Huybrechts I, Julia C, Kesse-Guyot E, Alles B, Galan P, Hercberg S, Pierre F, Deschasaux-Tanguy M, Touvier M. Dietary exposure to nitrites and nitrates in association with type 2 diabetes risk: Results from the NutriNet-Sante population-based cohort study. PLoS Med. 2023 Jan 17;20(1):e1004149. doi: 10.1371/journal.pmed.1004149. eCollection 2023 Jan. PMID 36649248
- [Derived] Debras C, Chazelas E, Sellem L, Porcher R, Druesne-Pecollo N, Esseddik Y, de Edelenyi FS, Agaesse C, De Sa A, Lutchia R, Fezeu LK, Julia C, Kesse-Guyot E, Alles B, Galan P, Hercberg S, Deschasaux-Tanguy M, Huybrechts I, Srour B, Touvier M. Artificial sweeteners and risk of cardiovascular diseases: results from the prospective NutriNet-Sante cohort. BMJ. 2022 Sep 7;378:e071204. doi: 10.1136/bmj-2022-071204. PMID 36638072
- [Derived] Peneau S, Benard M, Robert M, Alles B, Andreeva VA, Courtois F, Touvier M, Leys C, Bellisle F. Validation of the Flexible and Rigid Cognitive Restraint Scales in a General French Population. Int J Environ Res Public Health. 2022 Sep 30;19(19):12519. doi: 10.3390/ijerph191912519. PMID 36231817
- [Derived] Charreire H, Verdot C, Szabo de Edelenyi F, Deschasaux-Tanguy M, Srour B, Druesne-Pecollo N, Esseddik Y, Alles B, Baudry J, Deschamps V, Salanave B, Galan P, Hercberg S, Julia C, Kesse-Guyot E, Sapris Study Group, Bellicha A, Touvier M, Oppert JM. Correlates of Changes in Physical Activity and Sedentary Behaviors during the COVID-19 Lockdown in France: The NutriNet-Sante Cohort Study. Int J Environ Res Public Health. 2022 Sep 28;19(19):12370. doi: 10.3390/ijerph191912370. PMID 36231670
- [Derived] Kesse-Guyot E, Alles B, Brunin J, Fouillet H, Dussiot A, Mariotti F, Langevin B, Berthy F, Touvier M, Julia C, Hercberg S, Lairon D, Barbier C, Couturier C, Pointereau P, Baudry J. Nutritionally adequate and environmentally respectful diets are possible for different diet groups: an optimized study from the NutriNet-Sante cohort. Am J Clin Nutr. 2022 Dec 19;116(6):1621-1633. doi: 10.1093/ajcn/nqac253. PMID 36124645
- [Derived] Bellicha A, Wendeu-Foyet G, Coumoul X, Koual M, Pierre F, Gueraud F, Zelek L, Debras C, Srour B, Sellem L, Kesse-Guyot E, Julia C, Galan P, Hercberg S, Deschasaux-Tanguy M, Touvier M. Dietary exposure to acrylamide and breast cancer risk: results from the NutriNet-Sante cohort. Am J Clin Nutr. 2022 Oct 6;116(4):911-919. doi: 10.1093/ajcn/nqac167. PMID 36055962
- [Derived] Reuze A, Mejean C, Carrere M, Sirieix L, Druesne-Pecollo N, Peneau S, Touvier M, Hercberg S, Kesse-Guyot E, Alles B. Rebalancing meat and legume consumption: change-inducing food choice motives and associated individual characteristics in non-vegetarian adults. Int J Behav Nutr Phys Act. 2022 Sep 1;19(1):112. doi: 10.1186/s12966-022-01317-w. PMID 36050684
- [Derived] Berthy F, Brunin J, Alles B, Fezeu LK, Touvier M, Hercberg S, Galan P, Pointereau P, Lairon D, Baudry J, Kesse-Guyot E. Association between adherence to the EAT-Lancet diet and risk of cancer and cardiovascular outcomes in the prospective NutriNet-Sante cohort. Am J Clin Nutr. 2022 Oct 6;116(4):980-991. doi: 10.1093/ajcn/nqac208. PMID 35918246
- [Derived] Gisch UA, Robert M, Berlin N, Nebout A, Etile F, Teyssier S, Andreeva VA, Hercberg S, Touvier M, Peneau S. Mastery Is Associated With Weight Status, Food Intake, Snacking, and Eating Disorder Symptoms in the NutriNet-Sante Cohort Study. Front Nutr. 2022 May 25;9:871669. doi: 10.3389/fnut.2022.871669. eCollection 2022. PMID 35694168
- [Derived] Robert M, Shankland R, Bellicha A, Kesse-Guyot E, Deschasaux-Tanguy M, Andreeva VA, Srour B, Hercberg S, Touvier M, Leys C, Peneau S. Associations between Resilience and Food Intake Are Mediated by Emotional Eating in the NutriNet-Sante Study. J Nutr. 2022 Aug 9;152(8):1907-1915. doi: 10.1093/jn/nxac124. PMID 35641193
- [Derived] Rebouillat P, Vidal R, Cravedi JP, Taupier-Letage B, Debrauwer L, Gamet-Payrastre L, Guillou H, Touvier M, Fezeu LK, Hercberg S, Lairon D, Baudry J, Kesse-Guyot E. Prospective association between dietary pesticide exposure profiles and type 2 diabetes risk in the NutriNet-Sante cohort. Environ Health. 2022 May 25;21(1):57. doi: 10.1186/s12940-022-00862-y. PMID 35614475
- [Derived] Debras C, Chazelas E, Srour B, Druesne-Pecollo N, Esseddik Y, Szabo de Edelenyi F, Agaesse C, De Sa A, Lutchia R, Gigandet S, Huybrechts I, Julia C, Kesse-Guyot E, Alles B, Andreeva VA, Galan P, Hercberg S, Deschasaux-Tanguy M, Touvier M. Artificial sweeteners and cancer risk: Results from the NutriNet-Sante population-based cohort study. PLoS Med. 2022 Mar 24;19(3):e1003950. doi: 10.1371/journal.pmed.1003950. eCollection 2022 Mar. PMID 35324894
- [Derived] Deschasaux-Tanguy M, Srour B, Bourhis L, Arnault N, Druesne-Pecollo N, Esseddik Y, de Edelenyi FS, Allegre J, Alles B, Andreeva VA, Baudry J, Fezeu LK, Galan P, Julia C, Kesse-Guyot E, Peneau S, Hercberg S, Bajos N, Severi G, Zins M, de Lamballerie X, Carrat F, Touvier M; SAPRIS-SERO study group. Nutritional risk factors for SARS-CoV-2 infection: a prospective study within the NutriNet-Sante cohort. BMC Med. 2021 Nov 30;19(1):290. doi: 10.1186/s12916-021-02168-1. PMID 34844606
- [Derived] Debras C, Chazelas E, Srour B, Julia C, Kesse-Guyot E, Zelek L, Agaesse C, Druesne-Pecollo N, Andreeva VA, Galan P, Hercberg S, Latino-Martel P, Deschasaux-Tanguy M, Touvier M. Glycaemic index, glycaemic load and cancer risk: results from the prospective NutriNet-Sante cohort. Int J Epidemiol. 2022 Feb 18;51(1):250-264. doi: 10.1093/ije/dyab169. PMID 34491326
- [Derived] Carra MC, Fessi S, Detzen L, Darnaud C, Julia C, Hercberg S, Touvier M, Andreeva VA, Bouchard P. Self-reported periodontal health and incident hypertension: longitudinal evidence from the NutriNet-Sante e-cohort. J Hypertens. 2021 Dec 1;39(12):2422-2430. doi: 10.1097/HJH.0000000000002941. PMID 34261955
- [Derived] Schneider E, Sabate JM, Bouchoucha M, Debras C, Touvier M, Hercberg S, Benamouzig R, Buscail C, Julia C. FODMAP Consumption by Adults from the French Population-Based NutriNet-Sante Cohort. J Nutr. 2021 Oct 1;151(10):3180-3186. doi: 10.1093/jn/nxab207. PMID 34224572
- [Derived] Courtois F, Peneau S, Salanave B, Andreeva VA, Roland-Cachera MF, Touvier M, Galan P, Hercberg S, Fezeu LK. Trends in breastfeeding practices and mothers' experience in the French NutriNet-Sante cohort. Int Breastfeed J. 2021 Jul 2;16(1):50. doi: 10.1186/s13006-021-00397-x. PMID 34215307
- [Derived] Julia C, Leroy P, Adjibade M, Assmann KE, Touvier M, Hercberg S, Soler LG, Kesse-Guyot E. Public health potential of guidelines-based dietary scores for non-communicable diseases mortality prevention: simulation study using the Preventable Risk Integrated ModEl (PRIME) model. Public Health Nutr. 2021 Nov;24(16):5539-5549. doi: 10.1017/S1368980021002871. Epub 2021 Jul 2. PMID 34212836
- [Derived] Deschasaux-Tanguy M, Druesne-Pecollo N, Esseddik Y, de Edelenyi FS, Alles B, Andreeva VA, Baudry J, Charreire H, Deschamps V, Egnell M, Fezeu LK, Galan P, Julia C, Kesse-Guyot E, Latino-Martel P, Oppert JM, Peneau S, Verdot C, Hercberg S, Touvier M. Diet and physical activity during the coronavirus disease 2019 (COVID-19) lockdown (March-May 2020): results from the French NutriNet-Sante cohort study. Am J Clin Nutr. 2021 Apr 6;113(4):924-938. doi: 10.1093/ajcn/nqaa336. PMID 33675635
- [Derived] Egnell M, Boutron I, Peneau S, Ducrot P, Touvier M, Galan P, Buscail C, Porcher R, Ravaud P, Hercberg S, Kesse-Guyot E, Julia C. Randomised controlled trial in an experimental online supermarket testing the effects of front-of-pack nutrition labelling on food purchasing intentions in a low-income population. BMJ Open. 2021 Feb 8;11(2):e041196. doi: 10.1136/bmjopen-2020-041196. PMID 33558350
- [Derived] Mervant L, Tremblay-Franco M, Jamin EL, Kesse-Guyot E, Galan P, Martin JF, Gueraud F, Debrauwer L. Osmolality-based normalization enhances statistical discrimination of untargeted metabolomic urine analysis: results from a comparative study. Metabolomics. 2021 Jan 2;17(1):2. doi: 10.1007/s11306-020-01758-z. PMID 33389209
- [Derived] Kesse-Guyot E, Rebouillat P, Payrastre L, Alles B, Fezeu LK, Druesne-Pecollo N, Srour B, Bao W, Touvier M, Galan P, Hercberg S, Lairon D, Baudry J. Prospective association between organic food consumption and the risk of type 2 diabetes: findings from the NutriNet-Sante cohort study. Int J Behav Nutr Phys Act. 2020 Nov 9;17(1):136. doi: 10.1186/s12966-020-01038-y. PMID 33167995
- [Derived] Chazelas E, Debras C, Srour B, Fezeu LK, Julia C, Hercberg S, Deschasaux M, Touvier M. Sugary Drinks, Artificially-Sweetened Beverages, and Cardiovascular Disease in the NutriNet-Sante Cohort. J Am Coll Cardiol. 2020 Nov 3;76(18):2175-2177. doi: 10.1016/j.jacc.2020.08.075. No abstract available. PMID 33121725
- [Derived] Debras C, Chazelas E, Srour B, Kesse-Guyot E, Julia C, Zelek L, Agaesse C, Druesne-Pecollo N, Galan P, Hercberg S, Latino-Martel P, Deschasaux M, Touvier M. Total and added sugar intakes, sugar types, and cancer risk: results from the prospective NutriNet-Sante cohort. Am J Clin Nutr. 2020 Nov 11;112(5):1267-1279. doi: 10.1093/ajcn/nqaa246. PMID 32936868
- [Derived] Beslay M, Srour B, Mejean C, Alles B, Fiolet T, Debras C, Chazelas E, Deschasaux M, Wendeu-Foyet MG, Hercberg S, Galan P, Monteiro CA, Deschamps V, Calixto Andrade G, Kesse-Guyot E, Julia C, Touvier M. Ultra-processed food intake in association with BMI change and risk of overweight and obesity: A prospective analysis of the French NutriNet-Sante cohort. PLoS Med. 2020 Aug 27;17(8):e1003256. doi: 10.1371/journal.pmed.1003256. eCollection 2020 Aug. PMID 32853224
- [Derived] Rebouillat P, Vidal R, Cravedi JP, Taupier-Letage B, Debrauwer L, Gamet-Payrastre L, Touvier M, Hercberg S, Lairon D, Baudry J, Kesse-Guyot E. Estimated dietary pesticide exposure from plant-based foods using NMF-derived profiles in a large sample of French adults. Eur J Nutr. 2021 Apr;60(3):1475-1488. doi: 10.1007/s00394-020-02344-8. Epub 2020 Jul 30. PMID 32734347
- [Derived] Gehring J, Touvier M, Baudry J, Julia C, Buscail C, Srour B, Hercberg S, Peneau S, Kesse-Guyot E, Alles B. Consumption of Ultra-Processed Foods by Pesco-Vegetarians, Vegetarians, and Vegans: Associations with Duration and Age at Diet Initiation. J Nutr. 2021 Jan 4;151(1):120-131. doi: 10.1093/jn/nxaa196. PMID 32692345
- [Derived] Partula V, Deschasaux M, Druesne-Pecollo N, Latino-Martel P, Desmetz E, Chazelas E, Kesse-Guyot E, Julia C, Fezeu LK, Galan P, Hercberg S, Mondot S, Lantz O, Quintana-Murci L, Albert ML, Duffy D; Milieu Interieur Consortium; Srour B, Touvier M. Associations between consumption of dietary fibers and the risk of cardiovascular diseases, cancers, type 2 diabetes, and mortality in the prospective NutriNet-Sante cohort. Am J Clin Nutr. 2020 Jul 1;112(1):195-207. doi: 10.1093/ajcn/nqaa063. PMID 32369545
- [Derived] Chaltiel D, Julia C, Adjibade M, Touvier M, Hercberg S, Kesse-Guyot E. Adherence to the 2017 French dietary guidelines and adult weight gain: A cohort study. PLoS Med. 2019 Dec 30;16(12):e1003007. doi: 10.1371/journal.pmed.1003007. eCollection 2019 Dec. PMID 31887145
- [Derived] Srour B, Fezeu LK, Kesse-Guyot E, Alles B, Debras C, Druesne-Pecollo N, Chazelas E, Deschasaux M, Hercberg S, Galan P, Monteiro CA, Julia C, Touvier M. Ultraprocessed Food Consumption and Risk of Type 2 Diabetes Among Participants of the NutriNet-Sante Prospective Cohort. JAMA Intern Med. 2020 Feb 1;180(2):283-291. doi: 10.1001/jamainternmed.2019.5942. PMID 31841598
- [Derived] Seconda L, Egnell M, Julia C, Touvier M, Hercberg S, Pointereau P, Lairon D, Alles B, Kesse-Guyot E. Association between sustainable dietary patterns and body weight, overweight, and obesity risk in the NutriNet-Sante prospective cohort. Am J Clin Nutr. 2020 Jul 1;112(1):138-149. doi: 10.1093/ajcn/nqz259. PMID 31725157
- [Derived] Andrianasolo RM, Hercberg S, Kesse-Guyot E, Druesne-Pecollo N, Touvier M, Galan P, Varraso R. Association between dietary fibre intake and asthma (symptoms and control): results from the French national e-cohort NutriNet-Sante. Br J Nutr. 2019 Nov 14;122(9):1040-1051. doi: 10.1017/S0007114519001843. PMID 31340870
- [Derived] Chazelas E, Srour B, Desmetz E, Kesse-Guyot E, Julia C, Deschamps V, Druesne-Pecollo N, Galan P, Hercberg S, Latino-Martel P, Deschasaux M, Touvier M. Sugary drink consumption and risk of cancer: results from NutriNet-Sante prospective cohort. BMJ. 2019 Jul 10;366:l2408. doi: 10.1136/bmj.l2408. PMID 31292122
- [Derived] Adjibade M, Lemogne C, Touvier M, Hercberg S, Galan P, Assmann KE, Julia C, Kesse-Guyot E. The Inflammatory Potential of the Diet is Directly Associated with Incident Depressive Symptoms Among French Adults. J Nutr. 2019 Jul 1;149(7):1198-1207. doi: 10.1093/jn/nxz045. PMID 31152670
- [Derived] Srour B, Fezeu LK, Kesse-Guyot E, Alles B, Mejean C, Andrianasolo RM, Chazelas E, Deschasaux M, Hercberg S, Galan P, Monteiro CA, Julia C, Touvier M. Ultra-processed food intake and risk of cardiovascular disease: prospective cohort study (NutriNet-Sante). BMJ. 2019 May 29;365:l1451. doi: 10.1136/bmj.l1451. PMID 31142457
- [Derived] Benard M, Bellisle F, Kesse-Guyot E, Julia C, Andreeva VA, Etile F, Reach G, Dechelotte P, Tavolacci MP, Hercberg S, Peneau S. Impulsivity is associated with food intake, snacking, and eating disorders in a general population. Am J Clin Nutr. 2019 Jan 1;109(1):117-126. doi: 10.1093/ajcn/nqy255. PMID 30596882
- [Derived] Mejean C, Lampure A, Si Hassen W, Gojard S, Peneau S, Hercberg S, Castetbon K. Influence of food preparation behaviors on 5-year weight change and obesity risk in a French prospective cohort. Int J Behav Nutr Phys Act. 2018 Nov 26;15(1):120. doi: 10.1186/s12966-018-0747-4. PMID 30477513
- [Derived] Andreeva VA, Tavolacci MP, Galan P, Ladner J, Buscail C, Peneau S, Galmiche M, Hercberg S, Dechelotte P, Julia C. Sociodemographic correlates of eating disorder subtypes among men and women in France, with a focus on age. J Epidemiol Community Health. 2019 Jan;73(1):56-64. doi: 10.1136/jech-2018-210745. Epub 2018 Oct 9. PMID 30301763
- [Derived] Si Hassen W, Castetbon K, Peneau S, Tichit C, Nechba A, Lampure A, Bellisle F, Hercberg S, Mejean C. Socio-economic and demographic factors associated with snacking behavior in a large sample of French adults. Int J Behav Nutr Phys Act. 2018 Mar 15;15(1):25. doi: 10.1186/s12966-018-0655-7. PMID 29544552
- [Derived] Si Hassen W, Castetbon K, Tichit C, Peneau S, Nechba A, Ducrot P, Lampure A, Bellisle F, Hercberg S, Mejean C. Energy, nutrient and food content of snacks in French adults. Nutr J. 2018 Feb 27;17(1):33. doi: 10.1186/s12937-018-0336-z. PMID 29486784
- [Derived] Fiolet T, Srour B, Sellem L, Kesse-Guyot E, Alles B, Mejean C, Deschasaux M, Fassier P, Latino-Martel P, Beslay M, Hercberg S, Lavalette C, Monteiro CA, Julia C, Touvier M. Consumption of ultra-processed foods and cancer risk: results from NutriNet-Sante prospective cohort. BMJ. 2018 Feb 14;360:k322. doi: 10.1136/bmj.k322. PMID 29444771
- See also: PubMed abstract — https://www.ncbi.nlm.nih.gov/pubmed/20459807